CLINICAL TRIAL: NCT06916442
Title: A Single-Arm, Open-Label, Exploratory Study of Granzyme B-Targeted PET Imaging for Evaluating Tumor Response to Immunotherapy in Solid Tumors
Brief Title: Granzyme B-targeted PET Imaging Monitoring Tumor Responses to Immunotherapy
Acronym: GZMB_PET
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IITXM2024005; XKJS202026 (Other Grant/Funding Number: Discipline and Platform Development Fund of Zhongnan Hospital, Wuhan University); IITXM2024005 (Other Grant/Funding Number: Zhongnan Hospital of Wuhan University (Investigator-Initiated Trial Support Fund))
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: PET/CT; Solid Tumors, Adult; Solid Tumors, Advanced Solid Tumors
Keywords: Granzyme B; PET Imaging; Immunotherapy Response; Diagnostic Efficacy
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Immunotherapy Recipients with Malignant solid tumors: Participants: Adults (≥18 years) with histologically confirmed advanced solid tumors (e.g., NSCLC, HNSCC, et al) scheduled to receive immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1).
  Interventions:
  * Baseline: 18F-FDG PET/CT scan prior to immunotherapy initiation.
  * Post-treatment: Dual PET/CT imaging (GZMB-targeted and 18F-FDG) within one week after 1~2 cycles of immunotherapy.
  Objectives:
  * Compare the diagnostic accuracy of GZMB-targeted PET vs. 18F-FDG PET in distinguishing pseudoprogression (immune-related inflammatory response) from true progression.
  * Evaluate the ability of GZMB-targeted imaging to predict early immunotherapy response.
  Design: Single-arm observational study; PET parameters (SUVmax, tumor-to-background ratio, et al) will be correlated with clinical outcomes.
  Interventions: Diagnostic Test: PET/CT Imaging with GZMB-targeted tracer

INTERVENTIONS:
Diagnostic Test: PET/CT Imaging with GZMB-targeted tracer — Intravenous administration of GZMB-targeted tracer (150-200 MBq), followed by whole-body PET/CT scan 30~60 minutes post-injection.

SUMMARY:
Malignant solid tumors, characterized by their persistently high incidence and mortality rates, pose a significant threat to human health and life, imposing a substantial societal burden. Molecular imaging enables the non-invasive, in vivo visualization of tumorigenesis and progression at the molecular level. Compared to traditional morphology-based imaging techniques, molecular imaging provides more precise information for early tumor diagnosis, treatment efficacy assessment, and clinical disease management. 18F-FDG PET/CT imaging is currently the most widely used molecular imaging modality. However, under immunotherapy, FDG accumulates extensively in activated T cells, leading to increased false-positive evaluations. It fails to effectively distinguish metabolic hyperactivity between proliferative tumor cells (indicative of true progressive disease) and infiltrating immune cells (associated with pseudoprogression), thereby complicating the assessment of immunotherapy efficacy. Therefore, exploring novel molecular imaging probes with high specificity is of critical importance for patients undergoing tumor immunotherapy, as it can lead to more accurate evaluation of treatment efficacy. Granzyme B (GZMB), a serine protease released from cytoplasmic granules of cytotoxic T lymphocytes (CTLs) and natural killer (NK) cells, induces apoptosis in target cells, particularly tumor cells-a central mechanism of tumor immunotherapy. This makes GZMB a promising molecular target for evaluating immunotherapy efficacy. This study aims to assess tumor immunotherapy outcomes using GZMB-targeted PET imaging and compare its performance with 18F-FDG PET/CT. The goal is to achieve timely and accurate efficacy evaluation and longitudinal monitoring, identify potential beneficiaries, optimize clinical decision-making, and ultimately deliver personalized precision treatment to improve overall treatment outcomes.

DETAILED DESCRIPTION:
This investigator-initiated trial (IIT) aims to investigate the clinical utility of Granzyme B (GZMB)-targeted PET imaging for the early prediction of immunotherapy response in patients with malignant solid tumors. GZMB, a protease secreted by cytotoxic T lymphocytes, serves as a direct indicator of immune-mediated tumor killing activity. The GZMB-targeted tracer has demonstrated high target affinity and favorable pharmacokinetics in preclinical studies, showing potential to overcome the limitations of 18F-FDG PET in distinguishing between pseudoprogression and true progression.

In this prospective, single-arm observational study, patients with histologically confirmed malignant solid tumors (e.g., NSCLC, HNSCC, CRC, etc.) scheduled to receive immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1) will undergo baseline 18F-FDG PET/CT scans. Following 2~3 cycles of immunotherapy, they will undergo both GZMB-targeted PET/CT and 18F-FDG PET/CT scans within one week. PET parameters (SUVmax, SUVmean, tumor-to-background ratio) will be measured, calculated, and then correlated with pathologic response or objective response rate (ORR). The sensitivity, specificity, and accuracy of these parameters in monitoring tumor responses to immunotherapy will be analyzed. The diagnostic performance of both PET modalities will be compared. Additionally, this study will explore the correlations between PET parameters on GZMB-targeted PET imaging and the expression levels of GZMB and CD8+ in tumor tissue.

The study is funded by Zhongnan Hospital of Wuhan University. The results may establish GZMB-targeted PET imaging as a non-invasive tool for identifying patients likely to benefit from immunotherapy, thereby enabling the development of personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria

1. Voluntarily participate and sign the written informed consent form.
2. Aged 18 to 90 years (inclusive), regardless of gender.
3. Treatment-naïve patients with pathologically confirmed malignant solid tumors scheduled to receive immunotherapy.
4. Willing and able to adhere to scheduled visits, treatment plans, and laboratory tests.

Exclusion Criteria

1. Pregnant or lactating patients.
2. Patients with a known allergy to GZMB-targeted imaging agents or synthetic excipients.
3. Fasting blood glucose level exceeding 11.0 mmol/L prior to 18F-FDG administration.
4. Patients unable to undergo PET/CT imaging (e.g., inability to lie supine, claustrophobia, severe anxiety related to radiation exposure).
5. Patients with poor compliance or other factors deemed by the investigator to preclude participation in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants must voluntarily enroll and provide written informed consent, be aged 18 to 90 years (inclusive) regardless of gender, and have a pathologically confirmed diagnosis of treatment-naïve malignant solid tumors with planned immunotherapy. Additionally, participants must demonstrate willingness and ability to comply with scheduled clinical visits, adhere to prescribed treatment protocols, and complete required laboratory tests.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of Granzyme B targeted PET imaging monitoring tumor responses to immunotherapy | 4 years
  We will measure imaging parameters (SUVmax, SUVmean, tumor-to-background ratio), correlating with pathologic response or objective response rate (ORR). The sensitivity, specificity, and accuracy of these two PET/CT imaging modalities for early evaluation of immunotherapy response will be calculated/compared. This study will use pathological findings as the gold standard and clinical follow-up as a reference.

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou H, Wang Y, Xu H, Shen X, Zhang T, Zhou X, Zeng Y, Li K, Zhang L, Zhu H, Yang X, Li N, Yang Z, Liu Z. Noninvasive interrogation of CD8+ T cell effector function for monitoring early tumor responses to immunotherapy. J Clin Invest. 2022 Aug 15;132(16):e161065. doi: 10.1172/JCI161065. PMID 35788116